CLINICAL TRIAL: NCT05766722
Title: Feasibility of an Artificial Intelligence Phone Call for Post-operative Care Following Cataract Surgery in a Diverse Population
Brief Title: Feasibility of an Artificial Intelligence Phone Call After Cataract Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Uptown Eye Specialists (Other)
Responsible Party: Principal Investigator, Sohel Somani, Dr. Sohel Somani, clinical professor, Uptown Eye Specialists
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UptownEye3
Record Dates: First submitted 2022-08-17; First posted 2023-03-13 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Cataract
Keywords: Artificial Intelligence
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients 18 years old or older undergoing uncomplicated cataract surgery. (Experimental)
  Interventions: Device: DORA AI

INTERVENTIONS:
Device: DORA AI — Dora will phone patients on the day of cataract surgery (2 to 4 hours after discharge home) and again at postoperative week three. Dora calls made on the day of surgery will evaluate if the patient has any acute post-operative concerns like pain, and will prompt a postoperative day 1 visit if necessary. Calls to Dora at postoperative week three will result in either a follow-up to check refractive difficulties and/or confirmation of second eye surgery.

SUMMARY:
To analyze the evidence for clinical safety, usability, acceptability, satisfaction, appropriateness, and cost-effectiveness of Dora for recognizing patients who require additional in-person evaluation post cataract surgery. To assess Dora's sensitivity and specificity in cataract surgery management To determine what can be learnt to enhance AI technology in the field of ophthalmology especially when working with culturally diverse patients such as Punjabi and Chinese speaking patients.

DETAILED DESCRIPTION:
Background:

Cataract is defined as the degradation of the optical quality of the crystalline lens that affects vision and is the current leading cause of blindness worldwide. AI is set to revolutionize post-cataract surgery management by enhancing automation, increasing effectiveness, decreasing burdens placed on patients and the health care system. Ultimately, using AI-enabled automation could enhance patient management during and post cataract surgery.Cataract post-operative contact will be delivered by Dora agent, a natural language AI assistant.

Aim and objective:

Dora is a clinically safe, usable, appropriate, satisfactory and cost-effective AI technology for recognizing patients who require additional evaluation post cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are undergoing uncomplicated cataract surgery at a high volume surgical centre.

Exclusion Criteria:

* clinically significant complications during surgery that require more than the standard postop treatment or follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Dora is clinically safe | through study completion, an average of 4 weeks
  Clinical safety will be assessed using the comparison between Dora's clinical decision and the OT team's clinical decision.
Dora is usable | through study completion, an average of 4 weeks
  System usability scale will be used to assess usability of the technology. The scores are 0-100, a score above a 68 would be considered above average and anything below 68 is below average
Dora is clinically appropriate | through study completion, an average of 4 weeks
  System usability scale will be used to assess appropriateness of the technology. The scores are 0-100, a score above a 68 would be considered above average and anything below 68 is below average
Dora's clinical cost-effectiveness | through study completion, an average of 4 weeks
  Cost effectiveness will be assessed by comparing the cost of the system to the clinic specific costs (resources used and potential staff-hours) and patient specific costs (travel and time needed to be taken off from work)

SECONDARY OUTCOMES:
Multi-lingual capacity of AI technology | through study completion, an average of 4 weeks
  To determine what can be learnt to enhance AI technology in the field of ophthalmology especially when working with culturally diverse patients such as Punjabi and Chinese speaking patients by holding interviews from a randomly selected pool of applicants selected for an in-depth interview to better understand their experience with Dora such as challenges regarding communication and comprehension of the technology.

IPD SHARING:
Plan to Share IPD: Undecided